CLINICAL TRIAL: NCT06471244
Title: Development of Electroencephalography (EEG) and Magnetoencephalography (MEG) Source Reconstruction With Fast Multipole Method
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Worcester Polytechnic Institute (Other)
Collaborators: Technische Universität Ilmenau (Unknown); Max Planck Institute for Human Cognitive and Brain Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 24-0779
Record Dates: First submitted 2024-05-20; First posted 2024-06-24 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EEG/MEG data collection and processing with high density recording techniques (Experimental)
  Interventions: Other: Finger tapping; Other: Median nerve stimulation; Other: Speech processing

INTERVENTIONS:
Other: Finger tapping — The volunteer is tapping with his/her right hand index finger.
Other: Median nerve stimulation — Electrical pulses are applied at the wrist to the median nerve.
Other: Speech processing — German sentences are played to the volunteers and the volunteers have to fulfill a semantic task.

SUMMARY:
The goal of this clinical trial is to learn if an advanced 256 dry electrode EEG cap augmented with MEG readings and coupled with a new high-resolution fast brain modeling software gives a better EEG and MEG source localization in real time. The main questions it aims to answer are:

* Does the testbed better localize brain sources for finger movement?
* Does the testbed better localize brain sources for median nerve stimulation?
* Does the testbed better localize brain sources for speech processing?
* Researchers will compare the predicted cortical locations with MEG data and known anatomical locations of the neuronal generators.

Participants will:

* Undergo Magnetic Resonance Imaging (MRI) scans for brain and head model creation
* Undergo three different EEG tests
* Undergo three different MEG tests

DETAILED DESCRIPTION:
Magnetic Resonance Imaging (MRI) head/neck scans of 30 healthy subjects using the 7 Tesla Siemens Scanner will be performed at the Max Planck Institute for Human Cognitive and Brain Sciences, Leipzig Germany with 0.5/0.7 mm isotropic resolution, for both T1 and T2 imaging sequences. Construction of computational head models from the MRI data using FreeSurfer and Charm segmentation software packages will be performed at Worcester Polytechnic Institute.

On-skin voltage recordings will be done with 256 dry electrodes. Our EEG protocols will collect 240 trials per subject (3 runs of 80 trials each). German volunteers will be tapping with their right hand index finger. The corresponding neuronal generators are located in the M1INDEXFINGER/S1INDEXFINGER areas (primary motor/somatosensory cortex) at different latencies.

On-skin voltage recordings will be done with 256 dry electrodes. Our EEG protocols will collect 240 trials per subject (3 runs of 80 trials each). .Electrical stimuli over the median nerve at the right wrist will be delivered using brief transcutaneous pulses every 1.5 seconds. The task is to respond to each stimulus by pushing a button with the left-hand index finger. This generates EEG evoked responses in the S1HAND area (primary somatosensory cortex contralateral to the nerve stimuli), and the M1HAND area (primary motor cortex) at different latencies. The P20/N20 response peaking at about 20 ms is targeted, since at this latency its neuronal generators are well-known to be located in the posterior wall of the central sulcus in the Brodmann area 3b.

On-skin voltage recordings will be done with 256 dry electrodes. Our EEG protocols will collect 240 trials per subject (3 runs of 80 trials each). German sentences will be played to the volunteers and the volunteers have to fulfill a semantic task. This generates EEG evoked responses in the known areas of the Primary Auditory Cortex (PAC).

On-skin voltage recordings will be done with 256 dry electrodes. Our MEG protocols will collect 240 trials per subject (3 runs of 80 trials each). German volunteers will be tapping with their right hand index finger. The corresponding neuronal generators are located in the M1INDEXFINGER/S1INDEXFINGER areas (primary motor/somatosensory cortex) at different latencies.

On-skin voltage recordings will be done with 256 dry electrodes. Our MEG protocols will collect 240 trials per subject (3 runs of 80 trials each). Electrical stimuli over the median nerve at the right wrist will be delivered using brief transcutaneous pulses every 1.5 seconds. The task is to respond to each stimulus by pushing a button with the left-hand index finger. This generates MEG evoked responses in the S1HAND area (primary somatosensory cortex contralateral to the nerve stimuli), and the M1HAND area (primary motor cortex) at different latencies. The P20/N20 response peaking at about 20 ms is targeted, since at this latency its neuronal generators are well-known to be located in the posterior wall of the central sulcus in the Brodmann area 3b.

On-skin voltage recordings will be done with 256 dry electrodes. Our MEG protocols will collect 240 trials per subject (3 runs of 80 trials each). German sentences will be played to the volunteers and the volunteers have to fulfill a semantic task. This generates EEG evoked responses in the known areas of the Primary Auditory Cortex (PAC).

The main questions it aims to answer are:

Does the proposed high-resolution testbed better localize brain sources for finger movement?

Does the proposed high-resolution testbed better localize brain sources for median nerve stimulation?

Does the proposed high-resolution testbed better localize brain sources for speech processing?

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 and less than 66 years
* Normal hearing and (corrected) vision
* Able to understand and give informed consent

Exclusion Criteria:

* Cardiac pacemaker or pacemaker wires; neurostimulators; implanted pumps
* Metal in the body (rods, plates, screws, shrapnel, dentures, IUD) or metallic particles in the eye
* Surgical clips in the head or previous neurosurgery
* Any magnetic particles in the body
* Cochlear implants
* Prosthetic heart valves
* History of skull injury or defects
* Significant claustrophobia; Ménière's disease
* Pregnancy, breast feeding
* Neurological or psychiatric diagnoses or medications influencing brain function
* Current substance abuse (exception: concurrent nicotine use is allowed)
* Failure to perform the behavioral tasks or psychological evaluation tests
* Prisoners

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
MRI T1/T2 head/neck scans of 30 healthy subjects | 1 year
  Magnetic Resonance Imaging (MRI) head/neck scans of 30 healthy subjects using the 7 Tesla Siemens Scanner at the Max Planck Institute for Human Cognitive and Brain Sciences, Leipzig Germany with 0.5/0.7 mm isotropic resolution, for both T1 and T2 imaging sequencies. Construction of computational head models from the MRI data using FreeSurfer and Charm segmentation software packages.
EEG measurements of cortical activity in response to index finger tapping for 30 subjects | 1 year
  On-skin voltage recordings will be done with 256 dry electrodes. Our EEG protocols will collect 240 trials per subject (3 runs of 80 trials each). German volunteers will be tapping with their right hand index finger. The corresponding neuronal generators are located in the M1INDEXFINGER/S1INDEXFINGER areas (primary motor/somatosensory cortex) at different latencies.
EEG measurements of cortical activity in response to median nerve stimulation for 30 subjects | 1 year
  On-skin voltage recordings will be done with 256 dry electrodes. Our EEG protocols will collect 240 trials per subject (3 runs of 80 trials each). .Electrical stimuli over the median nerve at the right wrist will be delivered using brief transcutaneous pulses every 1.5 seconds. The task is to respond to each stimulus by pushing a button with the left-hand index finger. This generates EEG evoked responses in the S1HAND area (primary somatosensory cortex contralateral to the nerve stimuli), and the M1HAND area (primary motor cortex) at different latencies. The P20/N20 response peaking at about 20 ms is targeted, since at this latency its neuronal generators are well-known to be located in the posterior wall of the central sulcus in the Brodmann area 3b.
EEG measurements of cortical activity in response to auditory signals for 30 subjects | 1 year
  On-skin voltage recordings will be done with 256 dry electrodes. Our EEG protocols will collect 240 trials per subject (3 runs of 80 trials each). German sentences will be played to the volunteers and the volunteers have to fulfill a semantic task. This generates EEG evoked responses in the known areas of the Primary Auditory Cortex (PAC).
MEG measurements of cortical activity in response to index finger tapping for 30 subjects | through study completion, an average of 1 year
  On-skin voltage recordings will be done with 256 dry electrodes. Our MEG protocols will collect 240 trials per subject (3 runs of 80 trials each). German volunteers will be tapping with their right hand index finger. The corresponding neuronal generators are located in the M1INDEXFINGER/S1INDEXFINGER areas (primary motor/somatosensory cortex) at different latencies.
MEG measurements of cortical activity in response to median nerve stimulation for 30 subjects | through study completion, an average of 1 year
  On-skin voltage recordings will be done with 256 dry electrodes. Our MEG protocols will collect 240 trials per subject (3 runs of 80 trials each). Electrical stimuli over the median nerve at the right wrist will be delivered using brief transcutaneous pulses every 1.5 seconds. The task is to respond to each stimulus by pushing a button with the left-hand index finger. This generates MEG evoked responses in the S1HAND area (primary somatosensory cortex contralateral to the nerve stimuli), and the M1HAND area (primary motor cortex) at different latencies. The P20/N20 response peaking at about 20 ms is targeted, since at this latency its neuronal generators are well-known to be located in the posterior wall of the central sulcus in the Brodmann area 3b.
MEG measurements of cortical activity in response to auditory signals for 30 subjects | through study completion, an average of 1 year
  On-skin voltage recordings will be done with 256 dry electrodes. Our MEG protocols will collect 240 trials per subject (3 runs of 80 trials each). German sentences will be played to the volunteers and the volunteers have to fulfill a semantic task. This generates EEG evoked responses in the known areas of the Primary Auditory Cortex (PAC).

CONTACTS AND LOCATIONS:
Overall Officials: Sergey N Makaroff, PhD, Principal Investigator — Worcester Polytechnic Institute
Locations (2):
- Germany (2):
  - Technical University Ilmenau, Ilmenau
  - Max-Planck-Institut für Kognitions- und Neurowissenschaften [Cognitive and Neuroscience], Leipzig

IPD SHARING:
Plan to Share IPD: Yes
It is our firm intention to share our MRI/EEG/MEG datasets and resources with the broader neuroimaging and general scientific communities. The BEM-FMM computational package(s), along with the manual(s), application examples and supporting experimental data/human models, will be made available to interested researchers and collaborators, based on the widely accessible MATLAB platform for Windows and Linux following publication. Researchers with approved access to NIH-supported Scientific Data Repositories - the National Data Archive Database will be able to access raw experimental data from this project to enable sufficient independent validation efforts and to allow for replication of the research findings. The data will be available at The National Institute of Mental Health Data Archive (NDA) in accordance with the NIH Principles and Guidelines.
Supporting Information: Analytic Code
Time Frame: Data will become available as soon as practicable under the applicable study protocols.
Access Criteria: Access will be limited to qualified researchers through the NIMH Data Archive